CLINICAL TRIAL: NCT05767346
Title: A Phase 3, Multi-center, Randomized, Double-blind Trial to Evaluate the Efficacy and Safety of Aficamten Compared to Metoprolol in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: Phase 3 Trial to Evaluate the Efficacy and Safety of Aficamten Compared to Metoprolol Succinate in Adults With Symptomatic oHCM
Acronym: MAPLE-HCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CY 6032; 2023-504809-37-00 (Other: EU CTR Number)
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
Keywords: Obstructive Hypertrophic Cardiomyopathy; Aficamten; Metoprolol; oHCM; CK-3773274; CK-274; MAPLE-HCM; MAPLE; CY 6032
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aficamten up to 20 mg plus placebo for metoprolol (Experimental): Patients will receive doses of 5 mg, 10 mg, 15 mg or 20 mg of aficamten (CK-3773274) plus placebo for metoprolol succinate with dose levels guided by echocardiography assessments for up to 24 weeks.
  Interventions: Drug: Aficamten (CK-3773274) (5 mg, 10 mg, 15 mg and 20 mg); Drug: Placebo to match metoprolol succinate
- Metoprolol succinate up to 200 mg plus placebo for aficamten (Active Comparator): Patients will receive 50 mg, 100 mg, 150 mg or 200 mg of metoprolol succinate plus placebo for aficamten (CK-3773274) with dose levels guided by echocardiography and heart rate assessments for up to 24 weeks.
  Interventions: Drug: Placebo to match aficamten; Drug: Metoprolol succinate (50 mg, 100 mg, 150 mg and 200 mg)

INTERVENTIONS:
Drug: Aficamten (CK-3773274) (5 mg, 10 mg, 15 mg and 20 mg) — Aficamten (CK-3773274) tablets administered orally
  Arms: Aficamten up to 20 mg plus placebo for metoprolol
Drug: Placebo to match aficamten — Placebo for aficamten (CK-3773274) administered orally
  Arms: Metoprolol succinate up to 200 mg plus placebo for aficamten
Drug: Metoprolol succinate (50 mg, 100 mg, 150 mg and 200 mg) — Metoprolol succinate tablets administered orally
  Arms: Metoprolol succinate up to 200 mg plus placebo for aficamten
Drug: Placebo to match metoprolol succinate — Placebo for metoprolol succinate administered orally
  Arms: Aficamten up to 20 mg plus placebo for metoprolol

SUMMARY:
The purpose of this study is to compare the efficacy and safety of aficamten (CK-3773274) compared with metoprolol succinate in adults with symptomatic hypertrophic cardiomyopathy and left ventricular outflow tract obstruction

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet all the following criteria at screening may be included in the trial:

  * Males and females between 18 to 85 years of age, inclusive, at screening
  * Body mass index < 35 kg/m2
  * Diagnosed with oHCM per the following criteria by cardiac magnetic resonance imaging (CMR) or echocardiography -

    * Has left ventricular (LV) hypertrophy with non-dilated LV chamber in the absence of other cardiac disease and
    * Has an end-diastolic LV wall thickness as measured by the echocardiography core laboratory:

      1. ≥ 15 mm in one or more myocardial segments OR
      2. ≥ 13 mm in one or more wall segments and a known disease-causing gene mutation or positive family history of HCM
  * NYHA class II or III
  * Has a KCCQ-CSS score of ≤ 90 at screening
  * Has a screening echocardiogram with the following determined by the echocardiography core laboratory:

    * Resting LVOT-G > 30 mm Hg and/or post-Valsalva LVOT-G ≥ 50 mmHg at screening AND
    * LVEF ≥ 60%
  * Hemoglobin ≥ 10g/dL
  * Respiratory exchange ratio (RER) ≥ 1.05 and peak oxygen uptake (pVO2) < 100% predicted on the screening CPET per the core laboratory
  * Patients previously exposed to mavacamten are allowed to participate but must be off mavacamten for at least 8 weeks

Exclusion Criteria:

* Any of the following criteria will exclude potential participants from the trial:

  * Medical indication for either beta blocker or calcium-channel blockers prohibiting drug discontinuation other than oHCM
  * History of intolerance or medical contraindication to beta blocker therapy
  * Resting SBP of > 160 mmHg
  * Resting heart rate of > 100 bpm
  * Significant valvular heart disease

    1. Moderate-severe valvular aortic stenosis or fixed subaortic obstruction
    2. Mitral regurgitation not due to systolic anterior motion of the mitral valve (per Investigator judgment)
  * Known or suspected infiltrative, genetic or storage disorder causing cardiac hypertrophy that mimics oHCM (eg, Noonan syndrome, Fabry disease, amyloidosis)
  * History of LV systolic dysfunction (LVEF < 45%) or stress cardiomyopathy at any time during their clinical course
  * Inability to exercise on a treadmill or bicycle (eg, orthopedic limitations)
  * Documented room air oxygen saturation reading < 90% at screening
  * Planned septal reduction treatment that cannot be deferred during the trial period
  * History of septal reduction therapy (surgical myectomy or alcohol septal ablation) within 6 months of screening
  * History of paroxysmal or persistent atrial fibrillation or atrial flutter. Atrial flutter treated with radio frequency ablation without recurrence within the last 6 months prior to screening is allowed.
  * Current or recent (< 4 weeks) therapy with disopyramide
  * History of syncope, symptomatic ventricular arrhythmia, or sustained ventricular tachyarrhythmia with exercise within 6 months prior to screening
  * Has received prior treatment with aficamten or previously intolerant (reduced LVEF requiring permanent drug discontinuation) to mavacamten

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (pVO2) by cardiopulmonary exercise testing (CPET) | Baseline to Week 24
  Effect of aficamten compared with metoprolol succinate on exercise capacity in patients with symptomatic oHCM

SECONDARY OUTCOMES:
Proportion of patients with ≥1 class improvement in New York Heart Association (NYHA) Functional Class | Baseline to Week 24
  Effect of aficamten compared with metoprolol succinate on NYHA Functional Classification
Change in Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CSS) | Baseline to Week 24
  Effect of aficamten compared with metoprolol succinate on participant health status
Change in left ventricular mass index (LVMI) | Baseline to Week 24
  Effect of aficamten on mass of the heart as compared with metoprolol succinate
Change in left atrial volume index (LAVI) | Baseline to Week 24
  Effect of aficamten on size of the heart as compared with metoprolol succinate
Change from baseline values in NT-proBNP | Baseline to Week 24
  Effect of aficamten on NT-proBNP as compared with metoprolol succinate
Change in post-Valsalva LVOT-G | Baseline to Week 24
  Effect of aficamten on post-Valsalva LVOT-G as compared with metoprolol succinate

CONTACTS AND LOCATIONS:
Overall Officials: Scientific Leadership, Study Director — Cytokinetics
Locations (71):
- United States (28):
  - Alaska Heart and Vascular Institute, Anchorage, Alaska
  - Mayo Clinic, Phoenix, Arizona
  - UC San Diego Health - Sulpizio Cardiovascular Center, La Jolla, California
  - Cedars-Sinai Medical Center (Smidt Heart Institute), Los Angeles, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - AdventHealth, Orlando, Florida
  - Emory Clinic, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northwestern University, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Sanger Heart & Vascular Institute - HCM Clinic, Charlotte, North Carolina
  - Duke Health Center Arringdon, Morrisville, North Carolina
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Division of Heart Failure and Transplantation (Hospital of the University of Pennsylvania), Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Ascension Saint Thomas Heart West, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - CHI St. Luke's Health Baylor-St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Schar Heart and Vascular, Falls Church, Virginia
- Brazil (3):
  - Institutdo Danta Pazzanese, Ibirapuera, Ibirapuera
  - Instituto de Pesquisa Clinica de Campinas - IPECC, Campinas, São Paulo
  - lnstituto do Coracao do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
- Institut universitaire de cardiologie et de pneumonlogie de Quebec - Universite Laval, Québec, Canada
- China (6):
  - Xiangya Second Hospital of Central South University, Changsha
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhongshan Hospital Fudan University, Shanghai
  - Renmin Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital, Copenhagen
- France (6):
  - CHU La Timone, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Lariboisiere - APHP, Paris
  - Hopital Cardiologique Haut Leveque - CHU de Bordeaux, Pessac
  - CHU Pontchaillou, Rennes
  - Hopital Laennec - CHU de Nantes, Saint-Herblain
- Germany (3):
  - Charite-Universitatsmedizin Berlin - Campus Virchow Klinikum, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Jena, Jena
- Semmelweis Egyetem, Városmajori Szív- és Érgyógyászati Klinika, Budapest, Hungary
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Hadassah Hebrew Medical Center- Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
- AOU Careggi, Florence, Italy
- Erasmus Medical Center, Rotterdam, Netherlands
- Spain (8):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico Universitario Virgen Arrixaca, El Palmar
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Son Llatzer, Son Ferriol
- United Kingdom (6):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - Royal Brompton Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Oxford University Hospital NHS Trust - John Radcliffe Hospital - OCMR, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nassif ME, Garcia-Pavia P, Masri A, Merkely B, Pena-Pena ML, Barriales-Villa R, Bilen O, Burroughs M, Claggett BL, Costabel JP, de Barros Correia E, Dybro AM, Elliott P, Lakdawala NK, Lewis GD, Mann A, Maron MS, Miao ZM, Nair A, Poulsen SH, Reant P, Schulze PC, Solomon SD, Wang A, Sohn R, Berhane I, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Wohltman A, Fifer MA, Spertus JA; MAPLE-HCM Investigators. Effect of Aficamten vs Metoprolol on Patient-Reported Health Status in Obstructive Hypertrophic Cardiomyopathy. J Am Coll Cardiol. 2025 Nov 18:S0735-1097(25)10070-3. doi: 10.1016/j.jacc.2025.10.059. Online ahead of print. PMID 41493295
- [Derived] Wang A, Garcia-Pavia P, Masri A, Merkely B, Nassif ME, Pena-Pena ML, Barriales-Villa R, Bilen O, Burroughs M, Claggett BL, Costabel JP, de Barros Correia E, Dybro A, Elliott P, Hegde SM, Kulac IJ, Lakdawala NK, Lewis GD, Mann A, Nair A, Poulsen SH, Reant P, Schulze PC, Solomon SD, Sohn R, Berhane I, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Wohltman A, Fifer MA, Maron MS; MAPLE-HCM Investigators. Aficamten in Obstructive Hypertrophic Cardiomyopathy: A Multidomain, Patient-Level Analysis of the MAPLE-HCM Trial. J Am Coll Cardiol. 2025 Nov 18:S0735-1097(25)10068-5. doi: 10.1016/j.jacc.2025.10.057. Online ahead of print. PMID 41348072
- [Derived] Hegde SM, Wang X, Garcia-Pavia P, Getchevski S, Masri A, Merkely B, Nassif ME, Pena-Pena ML, Barriales-Villa R, Bilen O, Burroughs M, Claggett B, Costabel JP, Correia EB, Dybro AM, Elliott P, Lakdawala NK, Mann A, Maron MS, Nair A, Poulsen SH, Reant P, Schulze PC, Wang A, Sohn R, Berhane I, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Wohltman A, Fifer MA, Solomon SD; MAPLE-HCM Investigators. Effect of Aficamten Compared With Metoprolol on Echocardiographic Measures in Symptomatic Obstructive Hypertrophic Cardiomyopathy: MAPLE-HCM. J Am Coll Cardiol. 2025 Dec 16;86(24):2452-2467. doi: 10.1016/j.jacc.2025.08.022. Epub 2025 Aug 27. PMID 40932433
- [Derived] Garcia-Pavia P, Maron MS, Masri A, Merkely B, Nassif ME, Pena-Pena ML, Barriales-Villa R, Bilen O, Burroughs M, Claggett B, Costabel JP, Correia EB, Dybro AM, Elliott P, Hegde SM, Lakdawala NK, Lewis GD, Mann A, Miao ZM, Nair A, Poulsen SH, Reant P, Schulze PC, Solomon SD, Wang A, Sohn R, Berhane I, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Wohltman A, Fifer MA; MAPLE-HCM Investigators. Aficamten or Metoprolol Monotherapy for Obstructive Hypertrophic Cardiomyopathy. N Engl J Med. 2025 Sep 11;393(10):949-960. doi: 10.1056/NEJMoa2504654. Epub 2025 Aug 30. PMID 40888697
- [Derived] Garcia-Pavia P, Bilen O, Burroughs M, Costabel JP, de Barros Correia E, Dybro AM, Elliott P, Lakdawala NK, Mann A, Nair A, Nassif ME, Poulsen SH, Reant P, Schulze PC, Wang A, Berhane I, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Meng L, Sohn R, Wohltman A, Fifer MA; MAPLE-HCM Study Investigators. Aficamten vs Metoprolol for Obstructive Hypertrophic Cardiomyopathy: MAPLE-HCM Rationale, Study Design, and Baseline Characteristics. JACC Heart Fail. 2025 Feb;13(2):346-357. doi: 10.1016/j.jchf.2024.11.011. PMID 39909646